CLINICAL TRIAL: NCT01233687
Title: A Phase I/II Trial of AMG 102 and Erlotinib in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: AMG 102 and Erlotinib for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ahmad Tarhini (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-058
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Recurrent; progressive; advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — rilotumumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 102 and erlotinib (Experimental): Combination of AMG 102 and erlotinib
  Interventions: Drug: AMG 102 and erlotinib

INTERVENTIONS:
Drug: AMG 102 and erlotinib — Dose Level -2 Dose level -1 Dose Level 0 AMG 102 5 mg/kg 7.5 mg/kg 15 mg/kg Erlotinib 150 mg 150 mg 150 mg
  The first cohort of patients in the phase I portion will start at dose level 0 of AMG102.
  Other Names: Rilotumumab

SUMMARY:
This is a phase I/II study of erlotinib and AMG 102 in previously treated subjects with advanced NSCLC. Subjects will be enrolled with recurrent or progressive advanced stage NSCLC that has been treated with at least one and a maximum of two prior chemotherapy regimens. The Phase I part of the study will enroll 8-16 subjects with the Phase II part enrolling 21-45 subjects.

The Phase I part of the study is designed to determine how safest the combination of AMG 102 and erlotinib is and the recommended dose for the Phase II part. The Phase II part is to determine whether the combination of AMG102 and erlotinib works enough to warrant further interest in this combination.

DETAILED DESCRIPTION:
While modest improvements have been made in survival and quality of life in patients with advanced NSCLC there is a need to explore new agents and combinations with novel mechanisms of action in an effort to improve clinical outcomes in this patient population. The HGF/c-MET pathway inhibition is a promising novel target in NSCLC. Preclinical evidence support the combined targeting of EGFR and HGF/c-MET pathways in NSCLC as a strategy that may result in enhanced antitumor activity. Inhibition of both HGF/c-Met and EGFR pathways can be accomplished by utilizing the combination of AMG 102 and erlotinib in patients with advanced NSCLC. Therefore, we propose a safety and efficacy, phase I/II clinical trial of the combination in patients with previously treated, advanced NSCLC.

ELIGIBILITY:
Patients must have baseline evaluations performed prior to the first dose of study drug and must meet all inclusion and exclusion criteria. Results of all baseline evaluations, which assure that all inclusion and exclusion criteria have been satisfied, must be reviewed by a Physician Investigator prior to enrollment of that patient. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.

Inclusion Criteria:

* Patients with recurrent or progressive advanced stage Non-small cell lung cancer (NSCLC,no SCLC component) who have been treated with at least one and a maximum of two prior chemotherapy regimens for advanced NSCLC. Chemotherapy as part of initial potentially curative therapy (given as part of adjuvant or concomitant chemoradiotherapy) that was completed <1 year counts as 1 prior regimen. Prior erlotinib, other epidermal growth factor receptor (EGFR) TKIs or monoclonal antibodies targeting EGFR are not allowed.

NOTE: Chemotherapy as part of initial potentially curative therapy (given as part of adjuvant or concomitant chemoradiotherapy) that was completed one or more years prior to screening for this study does not count as a prior regimen.

If the tumor is refractory (progressed) after a prior chemotherapy regimen, then that regimen would count. If a prior chemotherapy regimen has been changed due to other reasons than disease progression (e.g. poor tolerance, allergic reaction), then it would not count as a separate prior regimen. A chemotherapy drug added for "maintenance" following disease stabilization or response to a chemotherapy regimen (in the absence of prior disease progression) does not count as a separate prior regimen.

NOTE: Pathology reports documenting the diagnosis of NSCLC are required to be reviewed by the screening physician investigator.

* Measurable disease (RECIST version 1.1) (for phase II part only).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 and life expectancy of ≥ 3 months.

NOTE: For the phase I part of the study, patients with ECOG Performance Status 2 will be excluded.

* Age ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Patients must meet the following laboratory criteria (within 14 days prior to study registration):

oHematology: Absolute neutrophil count (ANC) ≥ 1500/mm³ Platelets ≥ 100,000/mm³ Hemoglobin ≥ 9 g/dL International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits (WNL) of the institution oBiochemistry: Total Bilirubin within normal institutional limits. AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN), except if there is known hepatic metastasis, wherein transaminases may be ≤ 5 x institutional ULN.

Creatinine clearance 45 ml/min or higher calculated using the Cockcroft-Gault formula. Multiply the number by 0.85 if the patient is female.

* Patients must have fully recovered from the effects of any prior surgery, chemotherapy or radiation therapy. In the case of residual effects, these must be clinically stable, grade 1 or less in severity and do not meet other protocol exclusion criteria. A minimum time period of 3 weeks should elapse between the completion of radiation therapy for recurrent/metastatic disease and enrollment in the study. A minimum of 4 weeks should elapse between the completion of chemotherapy or any experimental therapy and enrollment in the study. A minimum of 4 weeks should elapse between prior major surgery (such as open biopsy or significant traumatic injury) and enrollment in the study. A minimum of 2 weeks should elapse between prior minor surgical procedures (such as chemotherapy infusion port placement or core visceral organ biopsy) and enrollment in the study.
* If patient has history of brain metastases, brain lesions should have been treated with surgery and/or radiation and be stable on repeat imaging and patients should be neurologically stable on a stable or tapering dose of corticosteroids.
* No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3-year disease-free interval.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method or abstain from sexual activity during the study and for 6 months after last study drug administration. Sexually active males and their female partners must agree to use two methods of accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study.
* All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required. This is due to the unknown effects of AMG102.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Patients who have mixed tumors with small-cell elements are ineligible.
* Pregnancy or lactation. All females of child-bearing potential must have negative serum or urine pregnancy tests within 7 days prior to starting study treatment.
* Prior treatment of NSCLC with EGFR TKIs or monoclonal antibodies targeting EGFR.
* A serious active infection (>grade 2) within 7 days of enrollment.
* A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Untreated brain metastases.
* A major surgical procedure or significant traumatic injury within 28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study per inclusion criterion 3.1. In addition, if a patient has not yet recovered from prior minor surgery (such as central venous access device or fine needle aspiration biopsy).
* Thrombosis or vascular ischemic events within the last twelve months, such as deep venous thrombosis, pulmonary embolism, transient ischemic attack, cerebral infarction, or myocardial infarction
* Concurrent or prior (within 7 days of enrollment) anticoagulation therapy, except for the use of low dose coumarin-type anticoagulants or low molecular weight heparin for prophylaxis against central venous catheter thrombosis
* Presence of peripheral edema > Grade 2 (CTCAE version 4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Phase I RP2D AMG 102 + Erlotinib
Arm/Group | AMG 102 + Erlotinib
Started | 7
Completed | 7
Not Completed | 0
Period: Phase II AMG 102 + Erlotinib
Arm/Group | AMG 102 + Erlotinib
Started | 49 (Includes 7 participants from Phase 1 part of study.)
Response-Evaluable | 45
Completed | 45
Not Completed | 4
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Experienced a Dose Limiting Toxicity
Description: Determination of the safety and recommended phase II dose of AMG 102 when combined with erlotinib for the treatment of patients with advanced, previously-treated NSCLC.
Time Frame: During first cycle of treatment (3 weeks)
Population: In the absence of DLTs among the first 7 pts treated, AMG 102 + Erlotinib (150 mg) daily (3 weeks) was declared the RP2D.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 7
percentage of participants | 0 [0 to 0]

2. Primary Outcome: Disease Control Rate (DCR)
Description: Using RECIST v1.1 criteria, DCR was determined by following equation: the number of complete response (CR) participants + the number of partial response (PR) participants + the number of stable disease (SD) participants / the number of complete response (CR) participants + the number of partial response (PR) participants + the number of stable disease (SD) participants + the number of progressive disease (PD) participants.
Time Frame: Six weeks from initiation of treatment with AMG 102 + Erlotinib
Population: All patients who who received at least one dose of AMG 102 and had post-treatment imaging studies for response evaluation using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria at six weeks (RESPONSE EVALUABLE)
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 45
percentage of patients | 60 [47 to 71]

3. Secondary Outcome: Objective Response Rate (ORR/Clinical Response)
Description: Using RECIST v1.1 criteria, ORR was determined by following equation: the number of partial response (PR) participants / the number of partial response (PR) participants + the number of stable disease (SD) participants + the number of progressive disease (PD) participants.
Time Frame: Up to 6 months
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 45
percentage of patients | 8.8 [0.4 to 18.4]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the start of treatment until first evidence of disease progression, death, or date of last contact. The (median) length of time that subjects with previously-treated advanced NSCLC, who were treated with the combination of AMG 102 and erlotinib, are both alive and free of disease progression as estimated by the Kaplan-Meier method. For participants not known to have died as of the data cut-off date and who did not have PD, the PFS date was censored at the last contact date (contacts considered in the determination of last progression free disease assessment).
Time Frame: Up to 24 months (after the first patient is accrued)
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 45
months | 2.6 [1.4 to 3.3]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was computed for all participants and is defined as the time between start of treatment and death. The (median) length of time in months that subjects with previously-treated advanced NSCLC, treated with the combination of AMG 102 and erlotinib, remain alive estimated by the Kaplan-Meier method.
Time Frame: Up to 24 months (after the first evaluable patient is accrued)
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AMG 102 + Erlotinib
Number analyzed (Participants) | 45
months | 6.6 [5.6 to 8.9]

ADVERSE EVENTS:
Groups:
- AMG 102 + Erlotinib: Serious and Non-Serious Adverse Events include the events considered at least possibly, probably or definitely related to study treatment.
  Non-Serious (Other) Adverse Events include those that occurred with a frequency of more than or equal to 5%.
Arm/Group | AMG 102 + Erlotinib
Serious Adverse Events (participants affected / at risk) | 18/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 + Erlotinib (N=45)
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 + Erlotinib (N=45)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 21
Vomiting (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 24
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 18
Platelet count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 7
Creatinine increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 10
Lymphocyte count decreased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 16
Anorexia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 20
Peripheral sensory neuropathy (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9
Rash acneiform (Skin and subcutaneous tissue disorders) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes